CLINICAL TRIAL: NCT02376400
Title: A Phase 1 Study to Evaluate the Safety, Tolerability and Immunogenicity of Heterologous Prime-Boost Regimens Using MVA-BN®-Filo and Ad26.ZEBOV Administered in Different Sequences and Schedules in Healthy Adults
Brief Title: A Study to Assess the Safety and Immunogenicity of Heterologous Prime-Boost Ebola Vaccine Regimens in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Crucell Holland BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR106459; VAC52150EBL1004 (Other: Crucell Holland BV)
Record Dates: First submitted 2015-01-26; First posted 2015-03-03 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Healthy
Keywords: Healthy; Ebola viruses; Ebola Viral Disease (EVD); Filoviruses; Monovalent vaccine; Human adenovirus serotype 26 (Ad26) expressing the Ebola virus Mayinga variant glycoprotein (Ad26.ZEBOV); Modified Vaccinia Virus Ankara - Bavarian Nordic Filo-vector (MVA-BN Filo); Safety; Immunogenicity

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Group 1 (Experimental): Participants will receive MVA-BN-filo/ Ad26.ZEBOV (Day 1 /Day 29) or Placebo (Day 1/Day 29).
  Interventions: Biological: MVA-BN-Filo; Biological: Ad26.ZEBOV; Biological: Placebo
- Group 2 (Experimental): Participants will receive MVA-BN-filo/Ad26.ZEBOV (Day 1 /Day 57) or placebo ( Day 1/Day 57).
  Interventions: Biological: MVA-BN-Filo; Biological: Ad26.ZEBOV; Biological: Placebo
- Group 3 (Experimental): Participants will receive Ad26.ZEBOV/ MVA-BN-filo (Day 1/Day 29) or placebo (Day 1/Day 29).
  Interventions: Biological: MVA-BN-Filo; Biological: Ad26.ZEBOV; Biological: Placebo
- Group 4 (Experimental): Participants will receive Ad26.ZEBOV/ MVA-BN-filo (Day 1/Day 57) or placebo (Day 1/Day 57).
  Interventions: Biological: MVA-BN-Filo; Biological: Ad26.ZEBOV; Biological: Placebo

INTERVENTIONS:
Biological: MVA-BN-Filo — One 0.5 milliliter (ml) intramuscular (IM) injection of 1*10^8, (50%Tissue Culture Infectious Dose [TCID50]) on Day 1, 29 or 57.
Biological: Ad26.ZEBOV — One 0.5 mL IM injection of 5*10^10 viral particles (vp) on Day 1, 29 or 57.
Biological: Placebo — One 0.5 mL IM injection of 0.9% saline on Day 1 and 29 or on Day 1 and 57.

SUMMARY:
The purpose of this study is to test the safety and immunogenicity of MVA-BN-Filo and Ad26.ZEBOV administered as heterologous prime-boost vaccine regimens in healthy adult participants.

DETAILED DESCRIPTION:
This is a randomized placebo-controlled, double-blind study evaluating the safety, tolerability and immunogenicity of MVA-BN-Filo and Ad26.ZEBOV administered in different sequences and schedules to healthy adult participants. The study consists of a screening period of up to 28 days, a vaccination period in which participants will be vaccinated at Baseline [Day 1] followed by a boost on Day 29 or 57 and a post-boost follow-up, until all participants have had their 21-day post-boost visit (Day 50 or Day 78). The participants who received active vaccine will enter a long-term follow-up. The total duration of the study will be about 1 year for participants who received vaccine and about 3 months for participants who received placebo. Immunogenicity and safety will be monitored during the study.

ELIGIBILITY:
Inclusion Criteria:

* Must be healthy on the basis of physical examination, medical history, and the investigator's clinical judgment
* Women of childbearing potential must have a negative serum beta-human chorionic gonadotropin pregnancy test at screening, a negative urine pregnancy test immediately prior to each study vaccine administration, and practice adequate birth control measures from 28 days before the prime vaccination until at least 3 months after the boost vaccination as specified in the study protocol. If not heterosexually active at screening, must agree to practice adequate birth control measures if they become heterosexually active during their participation in the study (from screening onwards until at least 3 months after the boost vaccination).
* Must be available and willing to participate for the duration of the study visits and follow-up, provide verifiable identification, and have a means to be contacted

Exclusion Criteria:

* Has been vaccinated with a candidate Ebola vaccine
* Has been diagnosed with Ebola disease or exposed to Ebola including travel to West Africa in the last 12 months. West Africa includes but is not limited to the countries of Guinea, Liberia, Mali, and Sierra Leone. Participants who anticipate traveling to epidemic Ebola areas before the start of the long-term follow-up period will also be excluded. During the long-term follow-up period, travel to epidemic Ebola areas is allowed but during this period sampling can only take place if participant has returned at least 1 month from the epidemic Ebola area to ensure the samples are not carrying the Ebola-virus
* Has received any Ad26- or MVA-based candidate vaccine in the past
* Known allergy or history of anaphylaxis or other serious adverse reactions to vaccines or vaccine products (including any of the constituents of the study vaccines), including known allergy to egg or aminoglycosides
* A woman who is pregnant or breast-feeding, or planning to become pregnant while enrolled in the study or within 3 months after the boost vaccination
* History of diabetes mellitus type 1 or type 2, including cases controlled with diet alone; thyroidectomy, or thyroid disease requiring medication during the last 12 months; uncontrolled hypertension as defined in the study protocol; or, major psychiatric illness and/or substance abuse problems during the past 12 months that in the opinion of the investigator would preclude participation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2015-04; Primary Completion 2015-12 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events | Up to 21 days post-boost (Day 50 for Groups 1 and 3 or Day 78 for Groups 2 and 4)
Number of Participants With Serious Adverse Events | Up to the end of long-term follow-up (day 360)
Number of Participants with Reactogenicity (that is, Solicited Local and Systemic Adverse Events) | 1 week after each study vaccine administration

SECONDARY OUTCOMES:
Immune Responses to the Study Vaccine Regimens as Measured by a Virus Neutralization Assay | Groups 1 and 3: Days 1 (pre-vaccination), 8, 29 (pre-vaccination), 36, 50, 113, 180, 240, and 360; Groups 2 and 4: Days 1 (pre-vaccination), 8, 29, 57 (pre-vaccination), 64, 78, 141, 180, 240, and 360)
Immune Responses to the Study Vaccine Regimens Measured by an Enzyme-linked Immunosorbent Assay (ELISA) | Groups 1 and 3: Days 1 (pre-vaccination), 8, 29 (pre-vaccination), 36, 50, 113, 180, 240, and 360; Groups 2 and 4: Days 1 (pre-vaccination), 8, 29, 57 (pre-vaccination), 64, 78, 141, 180, 240, and 360)
Immune Responses to the Study Vaccine Regimens as Measured by an Enzyme-linked Immunospot (ELIspot) Assay | Groups 1 and 3: Days 1 (pre-vaccination), 8, 29 (pre-vaccination), 36, 50, 113, 180, 240, and 360; Groups 2 and 4: Days 1 (pre-vaccination), 8, 29, 57 (pre-vaccination), 64, 78, 141, 180, 240, and 360)

CONTACTS AND LOCATIONS:
Overall Officials: Crucell Holland BV Clinical Trial, Study Director — Crucell Holland BV
Locations (2):
- Mwanza, Tanzania
- Entebbe, Uganda

REFERENCES:
- [Derived] Anywaine Z, Whitworth H, Kaleebu P, Praygod G, Shukarev G, Manno D, Kapiga S, Grosskurth H, Kalluvya S, Bockstal V, Anumendem D, Luhn K, Robinson C, Douoguih M, Watson-Jones D. Safety and Immunogenicity of a 2-Dose Heterologous Vaccination Regimen With Ad26.ZEBOV and MVA-BN-Filo Ebola Vaccines: 12-Month Data From a Phase 1 Randomized Clinical Trial in Uganda and Tanzania. J Infect Dis. 2019 Jun 5;220(1):46-56. doi: 10.1093/infdis/jiz070. PMID 30796818